CLINICAL TRIAL: NCT06621433
Title: Titanium-prepared Platelet Rich Fibrin Versus Connective Tissue Graft for Management of Type-2 Gingival Recession: a Randomized Controlled Clinical Trial
Brief Title: Titanium-prepared Platelet Rich Fibrin Versus Connective Tissue Graft for Management of Type-2 Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rizk Beshir (Other)
Responsible Party: Sponsor-Investigator, Rizk Beshir, MSc. candidate of periodontology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1/1-2023
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coronally advanced flap (CAF) in conjunction with titanium prepared PRF (Experimental)
  Interventions: Other: T-PRF with CAF
- CAF in conjunction with subepithelial connective tissue graft (SECTG) (Active Comparator)
  Interventions: Other: SECTG with CAF

INTERVENTIONS:
Other: T-PRF with CAF — Blood sample will be obtained from the patient, conveyed into a titanium tube and immediately centrifuged at 2700 rpm for 12 mins at room temperature using fixed angle centrifuge (PRF Process, Tangkula800-1, China). The fibrin clot will be collected and placed in the PRF compression device (PRF GRF box) and condensed to produce a uniform T-PRF membrane which will be inserted over the recession area and covered by the coronally advanced flap.
  Arms: Coronally advanced flap (CAF) in conjunction with titanium prepared PRF
Other: SECTG with CAF — Sub epithelial connective tissue graft will be obtained from the donor site (hard palate), placed into recipient site and secured by sutures, then covered by a coronally advanced flap.
  Arms: CAF in conjunction with subepithelial connective tissue graft (SECTG)

SUMMARY:
The aim of the study is to evaluate the effectiveness of using titanium prepared platelet rich fibrin with coronally advanced flap in the treatment of type-2 Cairo gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* Gingival recession type 2 according to Cairo et al (2011).
* Adequate amount of Attached Gingiva (AG) (2 mm≤ AG).
* Good oral hygiene (full mouth bleeding score and O'Leary index less than ≤10 % after complete phase I therapy)
* Clinically thick gingival biotype (1mm < gingival thickness).
* Anterior esthetic zone.

Exclusion Criteria:

* Patients with gingival recession types 1 and 3 according to Cairo et al.
* Inadequate amount of attached gingiva (AG < 2 mm).
* Uncooperative patients.
* Smoking more than 10 cigarettes per day.
* Patients with known systemic conditions or taking medications that may affect soft tissue healing.
* Pregnant and lactating women.
* Patients with parafunctional habits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Probing depth | up to 6 months
  The distance from the base of the pocket to the most apical point on the gingival margin will be measured using a periodontal probe.
Clinical attachment loss | up to 6 months
  Distance from the cement-enamel junction to the base of the periodontal pocket will be measured using a periodontal probe
Recession width (RW) | up to 6 months
  Recession width (W) measured at the widest point (it is the distance between the mesial gingival margin and the distal gingival margin of the tooth) using a periodontal probe
Recession height (RH) | up to 6 months
  It will be measured from the cementoenamel junction to the Gingival Margin (GM), parallel to the long axis of the tooth starting from the most apical point of the recession using a William's graduated periodontal probe
Width of keratinized gingiva (KT) | up to 6 months
  Width of keratinized gingiva will be measured as the distance from the gingival margin to the mucogingival junction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt